CLINICAL TRIAL: NCT06030323
Title: Validation and Testing of Artificial Intelligence Models to Measure Physical Activity in Patients Admitted to Hospital Following a Stroke
Brief Title: Validation of AI Models to Measure Physical Activity After a Stroke
Acronym: CaRRAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Peter Hartley, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A096458
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is not an interventional study. The study is classified as 'pre-clinical device development or performance testing'. The purpose of the study is to develop and validate the AI models using data collected from people affected by stroke in a hospital environment, to test the accuracy of the optimised models, and to ascertain patient preference for sensor location.

SUMMARY:
The research team are developing algorithms using artificial intelligence that use information collected by accelerometers to detect a person's position, such as whether an individual is lying, sitting, or standing, and the individual's movements, such as whether they are taking steps or standing up.

Sensor location will affect the accuracy of the model and acceptability of the method. The research team are therefore developing algorithms for four different locations.

The purpose of the research is for the development of the algorithms and check whether they accurately recognise different positions and movements in people whose movement is affected by a stroke, and by being in a hospital environment (e.g. using a profiling bed).

The research team plan to recruit between 34 and 50 participants who are admitted hospital due to having a stroke. After providing informed consent, participants will be asked to complete a one-off assessment with a member of the research team and a ward physiotherapist. Participants will be asked to wear the four sensors, and move through a series of postures, walk for up to six minutes, and stand as many times as they feel able in one minute.

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital with a diagnosis of an acute stroke.

Exclusion Criteria:

* unable to provide informed consent;
* receiving end-of-life care;
* the consultant in charge of their care disagrees with their inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute and sub-acute stroke inpatients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of AI models | Collected during hospitalisation (up to 12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom